CLINICAL TRIAL: NCT06651424
Title: Multicenter, Randomized, Double-blind, Parallel-group Controlled Nutritional Intervention Study to Evaluate the Effect of a Combination of Probiotic Strain on Postpartum Depression
Brief Title: Effect of Consuming a Combination of Probiotic Strains on Postpartum Depression
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: due to its evolution, evaluation, as well as other reasons shared and reviewed between the parties
Sponsor: Biosearch S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: P060
Record Dates: First submitted 2022-08-24; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Postpartum Depression
Keywords: Probiotics; Depression; Postpartum
MeSH Terms: conditions — Depression, Postpartum; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Pregnants will take 1 capsule with a combination of probiotics (no comercial) daily from the 32nd week gestation to the 4th week postpartum (approximately 12 weeks).
  Interventions: Dietary Supplement: Combination of Lactobacillus probiotics (no comercial)
- Control group (Placebo Comparator): Pregnants will take 1 capsule with maltodextrin daily from the 32nd week gestation to the 4th week postpartum (approximately 12 weeks).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Combination of Lactobacillus probiotics (no comercial) — Each participant will consume 1 capsule per day in one of the main meals without any restriction in the diet or in their life habits
  Arms: Experimental group
Dietary Supplement: Placebo — Each participant will consume 1 capsule per day in one of the main meals without any restriction in the diet or in their life habits
  Arms: Control group

SUMMARY:
The objective of this trial is to evaluate the effect of consuming a combination of Lactobacillus during the pregnancy and lactation period on the incidence of postpartum depression.

DETAILED DESCRIPTION:
The mood disorders such as postpartum depression have a very high incidence. There is a relationship between a woman's microbiota and the risk of postpartum depression.

The possibility of influencing the microbiota through probiotic treatments opens a door to the prevention and/or treatment of postpartum depression.

Therefore, the objective of this trial is to evaluate the effect of consuming a combination of Lactobacillus during the pregnancy and lactation period on the incidence of postpartum depression.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant who is between 28-32 weeks of gestation.
* Normal development of pregnancy.
* Singleton pregnancy.
* Score ≥12 scale Postpartum depression questionnaire Edinburgh.
* Pregnant who has the firm intention of breastfeeding her child for at least the first month.
* Sign the Informed Consent.

Exclusion Criteria:

* Have any breast pathology that makes it difficult or impossible to breastfeed.
* Consume other probiotic supplements during the study.
* History of serious mental disorders other than affective disorders, whether or not currently under pharmacological treatment.
* Low expectation of adherence to the study protocol.
* Pharmacological treatment incompatible with the study.
* Non-compliance with the study protocol.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant who is between 28-32 weeks of gestation.
Enrollment: 5 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Postpartum Depression | 12 weeks
  Edinburgh Postnatal Depression Scale (EPDS) (Score min=0; Max=30; The woman will be considered to have PPD if the Edinburgh Survey Scale score is ≥12)

SECONDARY OUTCOMES:
Changes in EPDS | 12 weeks
  Analysis of different scores on the scale EPDS
Incidence of anxiety | 12 weeks
  State-trait Anxiety Inventory (STAI-S) (score ≥40)
Changes in STAI-S | 12 weeks
  Analysis of different scores on the scale STAI-S
Assessment of pain during breastfeeding | 12 weeks
  McGill Pain Questionnaire adapted to breastfeeding
Cortisol in breast milk | 12 weeks
  2 samples (at week 1 postpartum and week 4 postpartum)
Cortisol in saliva | 12 weeks
  3 samples (at the beginning of the study, at week 38 of gestation and at week 4 postpartum)
Microbiota in breast milk | 12 weeks
  2 samples (at week 1 postpartum and week 4 postpartum)
Microbiota in mother's feces | 12 weeks
  2 samples (at the beginning of the study and at week 38 of gestation)
Comfort with breastfeeding | 12 weeks
  Survey on breastfeeding

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Blanco Rojo, PhD, Principal Investigator — Biosearch S.A.
Locations (3):
- Spain (3):
  - Hospital Universitario del Sureste (Arganda del Rey, Madrid), Arganda, Madrid
  - Clínica Luna de Brigantía (Vigo, Pontevedra), Vigo, Pontevedra
  - Centro de Salud Villacañas de Toledo, Villacañas, Toledo

IPD SHARING:
Plan to Share IPD: No